CLINICAL TRIAL: NCT00316420
Title: Phase I Trial of Gemcitabine and Capecitabine (Xeloda) in Patients With Advanced Pancreatic Carcinoma
Brief Title: Gemcitabine and Capecitabine in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Philip Gold, M.D., Swedish Medical Center, Swedish Cancer Insitute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TI027 PG/HK
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine (Xeloda) — 650 mg/m2 po bid Days 1-14 750 mg/m2 po bid Days 1-14 850 mg/m2 po bid Days 1-14 950 mg/m2 po bid Days 1-14
  Other Names: Xeloda
Drug: Gemcitabine — 750 mg/m2 IV Days 1 & 8 q 21 days
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to test the effectiveness and safety of the drug combination of gemcitabine and capecitabine (Xeloda) in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable pancreatic cancer
* No prior chemotherapy except radiation-sensitizing doses of 5-FU
* No radiotherapy less than 4 weeks prior to the start of the study

Exclusion Criteria:

* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-FU
* Moderate to severe renal impairment
* Uncontrolled diabetes
* Inability to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
MTD and DLT for the combination therapy of gemcitabine and capecitabine | January 2010

SECONDARY OUTCOMES:
Tumor Response | January 2010

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gold, MD, Principal Investigator — Swedish Medical Center Cancer Institute; Henry Kaplan, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (1):
- Swedish Medical Center Cancer Institute, Seattle, Washington, United States